CLINICAL TRIAL: NCT04444843
Title: A Multicenter Clinical Trial: Risk Factors of Chinese Kidney Transplant Recipients DSA Based on MPA Immunosuppressive Regimen
Brief Title: Risk Factors of Chinese Kidney Transplant Recipients DSA Based on MPA Immunosuppressive Regimen
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML40754
Record Dates: First submitted 2020-06-03; First posted 2020-06-24 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-04

CONDITIONS: Kidney Transplant Recipients
Keywords: kidney transplant recipients; Mycophenolate Mofetil Capsules; Acute Rejection; Cyclosporine; Delayed graft function; Tacrolimus; Mycophenolic Acid Area under the Curve
MeSH Terms: conditions — Delayed Graft Function | interventions — Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: To estimate the incidence of DSA formation during 12-months post-transplantation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mycophenolate Mofetil Capsules (Other): The dosage of mycophenolate mofetil (CellCept) will be decided by the investigator and should be adjusted according to clinical response or therapeutic drug monitoring. It is not allowed to switch to other MPAs. When MMF is discontinued but is not switched to other MPA, the patients will be followed until the end of study.
  Interventions: Drug: Mycophenolate Mofetil Capsules

INTERVENTIONS:
Drug: Mycophenolate Mofetil Capsules — Patients who received MMF+TAC+ Corticosteroids immunosuppressive regimen as first choice post transplantation
  Other Names: Other MPAs

SUMMARY:
THE INCIDENCE AND INFLUENTIAL FACTORS OF DSA IN CHINESE RENAL TRANSPLANT RECIPIENTS WITH MPA-BASED IMMUNOSUPPRESSIVE REGIMEN： A MULTI-CENTER CLINICAL STUDY (TIAIFOD STUDY)

Study procedure Investigators at participating centers will identify patients fulfilling inclusion criteria and do not violate any exclusion criteria. Informed consent will be obtained upon entry into the study according to national regulations. Patients will be enrolled into the study and clinical data of patient history will be collected. Clinical data will be collected prospectively up to a total period of 12 months.

DETAILED DESCRIPTION:
Medical history and Kidney transplantation This will include age at transplantation, gender, race, weight, height of both recipient and donor; Recipients: previous history ,BMI ,primary kidney disease including biopsy proven diagnosis (if present), historic dialysis，pregnancy history (female). Donor: the catalogue (DCD,DBD,DBCD), ECD or not，the cause of death, received CPR or not; zero biopsy results if done, ABO blood type match, HLA-MM, cold and warm ischemic time.

Clinical data at baseline and 12months follow up period:

Clinical assessments, laboratory, comorbidity, immunosuppressive therapy, and selected concomitant therapy (anti-hypertension anti-hyperlipidemics, anti-diabetics and drugs known to affect renal function) will be collected at transplant day（Day 0, visit 0）and 8 subsequent visits scheduled Day 3, Week1, Week2, Week 4，Week 12，Week 26，Week 40，Week 52 post transplantation. MPA-AUC, acute rejection episodes and graft loss will be collected at visits scheduled Day 3, Week 1，Week 2, Week 4，Week 12， Week 26(6 month)，Week 40，Week 52 (12 month) post transplantation. On day 3, MPA-AUC will be tested by full time sample (0h,0.5h,1h,2h,3h,4h,6h,8h,10h,12h post receiving MMF). LSS (0h, 0.5h, 2h post receiving MMF) will be used for testing MPA-AUC on other visits. PRA will be tested on week 4, week 12, week 26, week 52. If PRA is positive, DSA will be tested following once. All the PRA and DSA MFI and phenotype will be collected（including the clinical-drive test）.

Statistical analysis:

The primary endpoint in this study is the incidence of DSA formation in 12-months post-transplantation in Chinese kidney transplant recipients with MMF-based IS regimen. The proportion and its 95% CI will be provided.

The influential factors of DSA formation will be estimated using logistic regression including relevant influential factors, where the influential factors are defined as {age, gender of donor / recipients recipient: BMI, blood transfusion, previous AR （before DSA appears）, ECD , cold ischemia time, HLA-MM, Tac trough concentration, MPA-AUC, DGF, introduction therapy (including use or not and the drugs )}. .

The full MPA-AUC0-12h will be calculated using the trapezoidal rule. The calculated formula with Limited Sample Strategy (LSS) will be established to predict the MPA-AUC0-12h in the Chinese patients. Correlation coefficients will be calculated and multiple stepwise regression analysis will be used to determine the time points and best equation for evaluating MPA-AUC0-12h.

Estimates for the time-to-event variable(s), such as Overall Survival(OS), will be obtained by using the Kaplan-Meier (KM) approach together with associated 95% CI.

The other secondary endpoints will be summarized descriptively depended on the variable type. The comparison between patients with and without DSA-positive will be performed according to the variable type.

ELIGIBILITY:
Inclusion Criteria:

* Male or female kidney transplant recipients from 18 to 65 years of age (including 18 & 65 years old patients)
* Single organ and first kidney transplant recipients from donation after citizen's death
* Patients who received MMF+TAC+ Corticosteroids immunosuppressive regimen as first choice post transplantation
* Pre-transplant PRA is negative (0%)
* One serum pregnancy test with a sensitivity of at least 25mlU/Ml for patients of childbearing potential before enrolled. A second test should be performed 8-10 days later. Repeat pregnancy tests should be performed during routine follow-up visits. Results of all pregnancy tests should be discussed with the patient. Patients should be instructed to consult their physician immediately should pregnancy occur. For patients to be included in the study, negative result must be obtained. And highly effective contraception for women of childbearing potential. Contraception must be taken before beginning study drug therapy, during therapy and for 6 weeks after the last dose of study medication

Exclusion criteria:

* Patients who do not receive MMF
* Patients who are re-transplantation or multiple organ transplantation recipients
* Female patients who are pregnant or lactating
* Patients who have any form of substance abuse, psychological illness or any other condition, which, in the opinion of the investigator, may interfere with the patient's ability to understand the requirements of the study.
* Patients who would have received another investigational drug within 30 days preceding the enrollment, received prohibited immunosuppressant medications prior to transplant
* Patients who are using AZA, MTX, CTX or will use these drugs post-transplantation
* Known contraindications to TAC , corticosteroids, MMF
* Patients who have active peptic ulcer
* Patients who have severe cardiac or lung disease
* Patient who have active hepatica disease
* Patients who have a history of cancer, except successfully treated localized nonmelanocytic skin cancer
* Patients who would not be available for routine study visits or follow-up, or not being followed by an accredited laboratory.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-12-21 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of Donor specific antibody(DSA) formation during 12-months post-transplantation | 12-months
  the incidence of DSA formation during 12-months post-transplantation

SECONDARY OUTCOMES:
the incidence of DSA formation during 6-months post-transplantation | 6 months
  the incidence of DSA formation during 6-months post-transplantation
the influential factors of DSA formation | 12 months
  the influential factors of DSA formation
the association between DSA and MPA AUC | 12 months
  the association between DSA and MPA AUC
the calculation formula for MPA-AUC with ISS using multiple regression analysis | 12 months
  the calculation formula for MPA-AUC with ISS using multiple regression analysis
the proportion of patients experiencing Acute Rejection(AR), Biopsy proven acute rejection(BPAR), Antibody mediated rejection(ABMR) and the association with Donor specific antibody(DSA) | 12 months
  the proportion of patients experiencing AR, BPAR, ABMR and the association with DSA
the renal function (Calculated creatinine clearance) at 12 month and association with DSA | 12 months
  the renal function (Calculated creatinine clearance) at 12 month and association with DSA
the death-censored graft survival rate at 12 month post transplantation and association with Donor specific antibody(DSA) | 12 months
  the death-censored graft survival rate and association with Donor specific antibody(DSA)

CONTACTS AND LOCATIONS:
Overall Officials: Wujun Xue, Prof., Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital Xi'an Jiaotong University, Xi'an, Shaanxi, China

REFERENCES:
- [Result] Wolfe RA, Ashby VB, Milford EL, Ojo AO, Ettenger RE, Agodoa LY, Held PJ, Port FK. Comparison of mortality in all patients on dialysis, patients on dialysis awaiting transplantation, and recipients of a first cadaveric transplant. N Engl J Med. 1999 Dec 2;341(23):1725-30. doi: 10.1056/NEJM199912023412303. PMID 10580071
- [Result] Huang J, Millis JM, Mao Y, Millis MA, Sang X, Zhong S. Voluntary organ donation system adapted to Chinese cultural values and social reality. Liver Transpl. 2015 Apr;21(4):419-22. doi: 10.1002/lt.24069. Epub 2015 Feb 13. PMID 25545626
- [Result] Miettinen J, Perasaari J, Lauronen J, Qvist E, Valta H, Pakarinen M, Merenmies J, Jalanko H. Donor-specific HLA antibodies and graft function in children after renal transplantation. Pediatr Nephrol. 2012 Jun;27(6):1011-9. doi: 10.1007/s00467-012-2101-4. Epub 2011 Oct 13. PMID 21993970
- [Result] Meier-Kriesche HU, Schold JD, Srinivas TR, Kaplan B. Lack of improvement in renal allograft survival despite a marked decrease in acute rejection rates over the most recent era. Am J Transplant. 2004 Mar;4(3):378-83. doi: 10.1111/j.1600-6143.2004.00332.x. PMID 14961990
- [Result] Ginevri F, Nocera A, Comoli P, Innocente A, Cioni M, Parodi A, Fontana I, Magnasco A, Nocco A, Tagliamacco A, Sementa A, Ceriolo P, Ghio L, Zecca M, Cardillo M, Garibotto G, Ghiggeri GM, Poli F. Posttransplant de novo donor-specific hla antibodies identify pediatric kidney recipients at risk for late antibody-mediated rejection. Am J Transplant. 2012 Dec;12(12):3355-62. doi: 10.1111/j.1600-6143.2012.04251.x. Epub 2012 Sep 7. PMID 22959074
- [Result] Wiebe C, Gibson IW, Blydt-Hansen TD, Karpinski M, Ho J, Storsley LJ, Goldberg A, Birk PE, Rush DN, Nickerson PW. Evolution and clinical pathologic correlations of de novo donor-specific HLA antibody post kidney transplant. Am J Transplant. 2012 May;12(5):1157-67. doi: 10.1111/j.1600-6143.2012.04013.x. Epub 2012 Mar 19. PMID 22429309
- [Result] Everly MJ, Rebellato LM, Haisch CE, Ozawa M, Parker K, Briley KP, Catrou PG, Bolin P, Kendrick WT, Kendrick SA, Harland RC, Terasaki PI. Incidence and impact of de novo donor-specific alloantibody in primary renal allografts. Transplantation. 2013 Feb 15;95(3):410-7. doi: 10.1097/TP.0b013e31827d62e3. PMID 23380861
- [Result] Hidalgo LG, Campbell PM, Sis B, Einecke G, Mengel M, Chang J, Sellares J, Reeve J, Halloran PF. De novo donor-specific antibody at the time of kidney transplant biopsy associates with microvascular pathology and late graft failure. Am J Transplant. 2009 Nov;9(11):2532-41. doi: 10.1111/j.1600-6143.2009.02800.x. PMID 19843031
- [Result] Wiebe C, Gibson IW, Blydt-Hansen TD, Pochinco D, Birk PE, Ho J, Karpinski M, Goldberg A, Storsley L, Rush DN, Nickerson PW. Rates and determinants of progression to graft failure in kidney allograft recipients with de novo donor-specific antibody. Am J Transplant. 2015 Nov;15(11):2921-30. doi: 10.1111/ajt.13347. Epub 2015 Jun 10. PMID 26096305
- [Result] Cooper JE, Gralla J, Chan L, Wiseman AC. Clinical significance of post kidney transplant de novo DSA in otherwise stable grafts. Clin Transpl. 2011:359-64. PMID 22755431
- [Result] DeVos JM, Patel SJ, Burns KM, Dilioglou S, Gaber LW, Knight RJ, Gaber AO, Land GA. De novo donor specific antibodies and patient outcomes in renal transplantation. Clin Transpl. 2011:351-8. PMID 22755430
- [Result] de Kort H, Willicombe M, Brookes P, Dominy KM, Santos-Nunez E, Galliford JW, Chan K, Taube D, McLean AG, Cook HT, Roufosse C. Microcirculation inflammation associates with outcome in renal transplant patients with de novo donor-specific antibodies. Am J Transplant. 2013 Feb;13(2):485-92. doi: 10.1111/j.1600-6143.2012.04325.x. Epub 2012 Nov 21. PMID 23167441
- [Result] Sharma A, Lewis JR, Lim WH, Palmer S, Strippoli G, Chapman JR, Alexander SI, Craig JC, Wong G. Renal transplant outcomes and de novo donor-specific anti-human leukocyte antigen antibodies: a systematic review. Nephrol Dial Transplant. 2018 Aug 1;33(8):1472-1480. doi: 10.1093/ndt/gfy077. PMID 29660004
- [Result] O'Leary JG, Samaniego M, Barrio MC, Potena L, Zeevi A, Djamali A, Cozzi E. The Influence of Immunosuppressive Agents on the Risk of De Novo Donor-Specific HLA Antibody Production in Solid Organ Transplant Recipients. Transplantation. 2016 Jan;100(1):39-53. doi: 10.1097/TP.0000000000000869. PMID 26680372
- [Result] Pratschke J, Dragun D, Hauser IA, Horn S, Mueller TF, Schemmer P, Thaiss F. Immunological risk assessment: The key to individualized immunosuppression after kidney transplantation. Transplant Rev (Orlando). 2016 Apr;30(2):77-84. doi: 10.1016/j.trre.2016.02.002. Epub 2016 Feb 18. PMID 26965071
- [Result] Smith JM, Martz K, Blydt-Hansen TD. Pediatric kidney transplant practice patterns and outcome benchmarks, 1987-2010: a report of the North American Pediatric Renal Trials and Collaborative Studies. Pediatr Transplant. 2013 Mar;17(2):149-57. doi: 10.1111/petr.12034. Epub 2013 Jan 2. PMID 23281637
- [Result] Filler G, Lepage N. To what extent does the understanding of pharmacokinetics of mycophenolate mofetil influence its prescription. Pediatr Nephrol. 2004 Sep;19(9):962-5. doi: 10.1007/s00467-004-1571-4. Epub 2004 Jul 15. PMID 15257455
- [Result] Le Meur Y, Buchler M, Thierry A, Caillard S, Villemain F, Lavaud S, Etienne I, Westeel PF, Hurault de Ligny B, Rostaing L, Thervet E, Szelag JC, Rerolle JP, Rousseau A, Touchard G, Marquet P. Individualized mycophenolate mofetil dosing based on drug exposure significantly improves patient outcomes after renal transplantation. Am J Transplant. 2007 Nov;7(11):2496-503. doi: 10.1111/j.1600-6143.2007.01983.x. Epub 2007 Oct 1. PMID 17908276
- [Result] Tonshoff B, David-Neto E, Ettenger R, Filler G, van Gelder T, Goebel J, Kuypers DR, Tsai E, Vinks AA, Weber LT, Zimmerhackl LB. Pediatric aspects of therapeutic drug monitoring of mycophenolic acid in renal transplantation. Transplant Rev (Orlando). 2011 Apr;25(2):78-89. doi: 10.1016/j.trre.2011.01.001. Epub 2011 Mar 30. PMID 21454065
- [Result] Le Meur Y, Borrows R, Pescovitz MD, Budde K, Grinyo J, Bloom R, Gaston R, Walker RG, Kuypers D, van Gelder T, Kiberd B. Therapeutic drug monitoring of mycophenolates in kidney transplantation: report of The Transplantation Society consensus meeting. Transplant Rev (Orlando). 2011 Apr;25(2):58-64. doi: 10.1016/j.trre.2011.01.002. Epub 2011 Mar 30. No abstract available. PMID 21454067
- [Result] Pawinski T, Hale M, Korecka M, Fitzsimmons WE, Shaw LM. Limited sampling strategy for the estimation of mycophenolic acid area under the curve in adult renal transplant patients treated with concomitant tacrolimus. Clin Chem. 2002 Sep;48(9):1497-504. PMID 12194926
- [Result] Magee JC, Krishnan SM, Benfield MR, Hsu DT, Shneider BL. Pediatric transplantation in the United States, 1997-2006. Am J Transplant. 2008 Apr;8(4 Pt 2):935-45. doi: 10.1111/j.1600-6143.2008.02172.x. PMID 18336697
- [Result] Chen B, Gu Z, Chen H, Zhang W, Fen X, Cai W, Fan Q. Establishment of high-performance liquid chromatography and enzyme multiplied immunoassay technology methods for determination of free mycophenolic acid and its application in Chinese liver transplant recipients. Ther Drug Monit. 2010 Oct;32(5):653-60. doi: 10.1097/FTD.0b013e3181f01397. PMID 20814351
- [Result] Filler G, Todorova EK, Bax K, Alvarez-Elias AC, Huang SH, Kobrzynski MC. Minimum mycophenolic acid levels are associated with donor-specific antibody formation. Pediatr Transplant. 2016 Feb;20(1):34-8. doi: 10.1111/petr.12637. Epub 2015 Nov 21. PMID 26589470
- [Result] Metzger RA, Delmonico FL, Feng S, Port FK, Wynn JJ, Merion RM. Expanded criteria donors for kidney transplantation. Am J Transplant. 2003;3 Suppl 4:114-25. doi: 10.1034/j.1600-6143.3.s4.11.x. No abstract available. PMID 12694055
- [Result] Mallon DH, Summers DM, Bradley JA, Pettigrew GJ. Defining delayed graft function after renal transplantation: simplest is best. Transplantation. 2013 Nov 27;96(10):885-9. doi: 10.1097/TP.0b013e3182a19348. PMID 24056620
- [Result] Czyzewski L, Wyzgal J, Czyzewska E, Kurowski A, Sierdzinski J, Labus A, Truszewski Z, Szarpak L. Performance of the MDRD, CKD-EPI, and Cockcroft-Gault Formulas in Relation to Nutritional Status in Stable Renal Transplant Recipients. Transplant Proc. 2016 Jun;48(5):1494-7. doi: 10.1016/j.transproceed.2016.01.083. PMID 27496434
- [Result] Malheiro J, Tafulo S, Dias L, Martins LS, Fonseca I, Beirao I, Castro-Henriques A, Cabrita A. Analysis of preformed donor-specific anti-HLA antibodies characteristics for prediction of antibody-mediated rejection in kidney transplantation. Transpl Immunol. 2015 Mar;32(2):66-71. doi: 10.1016/j.trim.2015.01.002. Epub 2015 Feb 7. PMID 25661873
- [Result] Haas M, Loupy A, Lefaucheur C, Roufosse C, Glotz D, Seron D, Nankivell BJ, Halloran PF, Colvin RB, Akalin E, Alachkar N, Bagnasco S, Bouatou Y, Becker JU, Cornell LD, Duong van Huyen JP, Gibson IW, Kraus ES, Mannon RB, Naesens M, Nickeleit V, Nickerson P, Segev DL, Singh HK, Stegall M, Randhawa P, Racusen L, Solez K, Mengel M. The Banff 2017 Kidney Meeting Report: Revised diagnostic criteria for chronic active T cell-mediated rejection, antibody-mediated rejection, and prospects for integrative endpoints for next-generation clinical trials. Am J Transplant. 2018 Feb;18(2):293-307. doi: 10.1111/ajt.14625. Epub 2018 Jan 21. PMID 29243394
- [Result] van Gelder T, Silva HT, de Fijter JW, Budde K, Kuypers D, Tyden G, Lohmus A, Sommerer C, Hartmann A, Le Meur Y, Oellerich M, Holt DW, Tonshoff B, Keown P, Campbell S, Mamelok RD. Comparing mycophenolate mofetil regimens for de novo renal transplant recipients: the fixed-dose concentration-controlled trial. Transplantation. 2008 Oct 27;86(8):1043-51. doi: 10.1097/TP.0b013e318186f98a. PMID 18946341